CLINICAL TRIAL: NCT06562478
Title: Effects of Zazen Meditation on Physiological and Psychological Aspects in Patients With Acute Myocardial Infarction - Randomized Clinical Trial
Brief Title: Effects of Zazen Meditation in Patients With Acute Myocardial Infarction - Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2019-0506
Record Dates: First submitted 2024-04-26; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Heart Rate Variability; Acute Myocardial Infarction
Keywords: Myocardial Infarction; heart rate variability
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Intervention (Active Comparator): Aspects of Zazen will be addressed. In the first session, the practice will be conducted for a duration of 5 minutes. In the second session, the duration will be extended to 10 minutes, aiming to provide adaptation for the participants. In the third session, the practice will last for 15 minutes, during which heart rate variability will be measured using the Polar H10 chest strap and the Elite HRV mobile app, both before and after the practice, to assess acute effects. At the end of the 24 sessions, the chronic effects of the practices will be evaluated in the same manner.
  Interventions: Behavioral: Zazen Meditation
- Documentary Control (Active Comparator): Neutral documentary on quality of life, for 30 minutes twice a week. Both groups will undergo intervention twice a week for 3 months, totaling 24 sessions. In the third session, heart rate variability assessment will be conducted to observe the acute effects of the method.
  Interventions: Behavioral: Zazen Meditation

INTERVENTIONS:
Behavioral: Zazen Meditation — The sessions will last a maximum of 40 minutes in total, comprising 10 minutes of introduction with general practice instructions, followed by 15 minutes of Zazen meditation practice. The final 15 minutes will be allocated for participants to provide feedback on the session.

SUMMARY:
Introduction: Coronary Artery Disease (CAD) remains the leading cause of death in Brazil, with literature indicating that in patients post-acute myocardial infarction, reduced Heart Rate Variability (HRV) has been established as a risk factor. One of the studied practices to aid in rehabilitation is meditation, believed to alter physiological aspects related to stress such as respiratory rate, oxygen consumption, carbon dioxide production, and systolic blood pressure, suggesting a better sympathetic-vagal balance. Objective: To assess the effects of Zazen meditation practice on heart rate variability in patients with recent acute and chronic myocardial infarction. Methodology: Randomized Clinical Trial. Chronic assessments will include: HRV with Polar H10 heart rate monitor, Quality of Life assessment with SF36 Quality of Life and Health questionnaire, Spiritual assessment with WHOQOL SR Spirituality, Religiosity, and Personal Beliefs questionnaire, Biochemical Parameters with ultra-sensitive PCR and cortisol, Ventricular Ejection Fraction (VEF), and 6-minute Walk Test (6MWT). Acute assessments will include: HRV with Polar H10 heart rate monitor, before and after a meditation session, in time and frequency domains. Sample size calculation was performed using Winpepi software version 11.43, with a power of 80% and significance level of 5%, determining a sample of 44 individuals. For intra-group differences analysis, ANOVA for repeated measures and/or its non-parametric counterpart, Friedman Test, will be used. For proportion analysis and comparison, Chi-square Test will be used. Expected Results: It is expected that the findings will contribute to a better understanding of the potential benefits that a meditation intervention may bring to patients who have experienced acute myocardial infarction.

DETAILED DESCRIPTION:
Chronic Study: The chronic effects of meditation practice will be evaluated at the beginning of the study and after 12 weeks of intervention. All study participants, regardless of group, will be invited to attend an initial conversation where all study procedures and assessments will be explained. Any questions will be clarified, and necessary explanations will be provided. After signing the Informed Consent Form (ICF), evaluations related to the chronic effects of meditation will be conducted, including the administration of specific questionnaires, resting HRV assessment, HRV assessment after the Stroop Test, 6-minute Walk Test (6MWT), and blood collection. Once all evaluations are completed, participants will be cleared to proceed with the study and begin the sessions.

At the end of each meditation session, participants will be invited to have tea with the researchers to report any comforts or discomforts experienced during the intervention. After completing the chronic study, i.e., after the 24 sessions, participants will repeat the same initial assessments conducted at the beginning of the study.

Acute Study: The acute study will occur simultaneously with the chronic study, as part of the Randomized Clinical Trial. Acute effects will be evaluated during the third intervention session in both groups, i.e., in the meditation and documentary sessions. On this day, participants must arrive 40 minutes before the session begins for the placement of the Polar H10 and to receive further instructions to ensure the quality of the assessment. Participants will remain at rest for ten minutes while being monitored, and after the protocol is completed, HRV will be recorded for the 5 minutes before the start of the session and for the 5 minutes after the session ends.

ELIGIBILITY:
Inclusion Criteria:

* Recent acute myocardial infarction
* Both sexes
* >18 years old
* Availability to attend the hospital at least twice a week during the study period
* Agree to the study and sign the Free and Informed Consent Form.

Exclusion Criteria:

* Unstable angina
* Extensive residual myocardial ischemia (at rest or on exertion)
* Inadequate blood pressure response during exercise
* Congestive heart failure class III or IV
* Severe lung disease
* Difficulty or inability to walk
* Pacemaker
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability | up to 12 weeks
  Assessed using the Polar H10 heart rate monitor, before and after a meditation session to evaluate acute effects, and before and after 24 sessions to evaluate chronic effects.

SECONDARY OUTCOMES:
Assessment of Quality of Life through the Quality of Life and Health Questionnaire | up to 12 weeks
  Quality of Life and Health
Assessment of Spirituality through the Spirituality, Religiosity, and Personal Beliefs | up to 12 weeks
  Questionnaire
Blood Tests | up to 12 weeks
  Ultra-sensitive C-reactive protein and cortisol.
Echocardiography | up to 12 weeks
  Ejection Fraction
Six-Minute Walk Test | up to 12 weeks
  Functional Capacity

CONTACTS AND LOCATIONS:
Overall Officials: Rosane M Nery, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No